CLINICAL TRIAL: NCT05117684
Title: To Compare "Balloon Occluded Thrombolysis" With "Conventional Catheter Directed Thrombolysis" in Thrombotically Occluded DIPSS Stent in Patients of Budd- Chiari Syndrome.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Budd-Chiari-01
Record Dates: First submitted 2021-10-30; First posted 2021-11-11 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Budd-Chiari Syndrome
MeSH Terms: conditions — Budd-Chiari Syndrome | interventions — Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novel: Balloon- Occlusion thrombolysis was done in adjunct to thrombus maceration, balloon sweeping and thrombosuction.
  Interventions: Procedure: Novel
- Conventional: Continuous catheter directed thrombolysis (Continuous urokinase infusion) was done along with thrombus maceration, balloon sweeping and thrombosuction.
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Novel — Balloon- Occlusion thrombolysis was done in adjunct to thrombus maceration, balloon sweeping and thrombosuction.
  Groups: Novel
Procedure: Conventional — Continuous catheter directed thrombolysis (Continuous urokinase infusion) was done along with thrombus maceration, balloon sweeping and thrombosuction.
  Groups: Conventional

SUMMARY:
DIPSS has become a widely accepted treatment for complications of portal hypertension. Shunt or hepatic vein stenosis are common short and mid term complications of the procedure. When identified early, shunt stenosis or occlusion may be treated before recurrence of the symptoms for which DIPSS was done at the first place. Present day endovascular DIPSS revision techniques have significantly improved the primary assisted patency rates.

The purpose of this study is to understand the newer technique of Combined balloon occlusion thrombolysis and intra stent balloon sweeping being practiced at our institute and compare it with the widely used conventional thrombolytic methods.

DETAILED DESCRIPTION:
Primary objective:

1. To study the outcome of combined technique of Balloon occluded thrombolysis, Balloon sweeping and maceration of thrombus in Blocked DIPSS stent and compare it with Conventional catheter directed thrombolysis and angioplasty.

   Secondary objective:
2. Study DIPSS stent patency and re-occlusion rates at 1 month followup

Methodology:

Study population: Patients with Budd -Chiari syndrome who underwent DIPSS revision till February 2021

Study design: Single center retrospective cohort study

Study period: 1year

Sample size: All eligible patients according to inclusion and exclusion criteria who underwent TIPS/DIPS revision will be included in thestudy.

Intervention: DIPSS Revision

Monitoring andassessment:

The following parameters to be evaluated over a period at least 1 month after DIPSS revision and compare with pre revisionvalues

Clinical parameters:

Status of ascites Urine output Recurrence of UGI/LGI bleed

Laboratory parameters:

ALBI Score,LFT, KFT

DOPPLER PARAMETERS:

Mid stent velocity, velocity at hepatic venous end Main portal vein velocity Direction of flow in intrahepatic portal vein branches

Stopping rule: Not applicable.

Expected outcome of the project: Balloon Occluded thrombolytic infusion alongwith intratsent balloon sweeping gives faster and better patency as compared to conventional pharmaco-mechanicalthrombolytic methods

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Budd- Chiari syndrome who underwent DIPSS revision for blocked stent till February 2021

Exclusion Criteria:

1. Patients who underwent DIPSS revision more than one time using both the techniques were excluded.
2. Failure to cannulate existing shunt.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Budd -Chiari syndrome who underwent DIPSS revision till February 2021
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Compare the rate of re-stenting between the two groups | Day 0
Compare the mean total dose of thrombolytic drug administered between the two groups | Day 0

SECONDARY OUTCOMES:
Study DIPSS stent patency and re-occlusion rates at 1 month followup. | 1 month
To compare the length of hospital stay between two groups | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided